CLINICAL TRIAL: NCT01909830
Title: A Phase II Study to Evaluate Activity and Toxicity of Gemcitabine in Combination With Pemetrexed Long Term Infusion in the Treatment of Pretreated Metastatic Colorectal Cancer Patients
Brief Title: Gemcitabine in Combination With Pemetrexed Long Term Infusion in the Treatment of Pretreated Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST153.03; 2010-019841-25 (EudraCT Number)
Record Dates: First submitted 2013-06-19; First posted 2013-07-29 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal Cancer Metastatic; pretreated
MeSH Terms: interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A : Gemcitabine + Pemetrexed (Experimental): Arm A : Gemcitabine: 1000 mg/m2 by intravenous infusion over an exact period of 30' (preferably by a pump to guarantee a constant speed of infusion) on day 3 of each cycle repeated every 14 days.
  Pemetrexed: 150 mg/m2 by intravenous continuous infusion over an exact period of 8h on day 1 of each cycle repeated every 14 days.
  Interventions: Drug: Arm A : Gemcitabine + Pemetrexed

INTERVENTIONS:
Drug: Arm A : Gemcitabine + Pemetrexed — Gemcitabine: 1000 mg/m2 by intravenous infusion over an exact period of 30' (preferably by a pump to guarantee a constant speed of infusion) on day 3 of each cycle repeated every 14 days.
  Pemetrexed: 150 mg/m2 by intravenous continuous infusion over an exact period of 8h on day 1 of each cycle repeated every 14 days.
  Other Names: Gemcitabine; Pemetrexed

SUMMARY:
Study Design:

Multicenter, non randomized, open label phase II study designed to evaluate the efficacy and safety of Gemcitabine/Pemetrexed combination.

Enrollment period: 18 months. Treatment period: maximum for 24 weeks for each patient (12 cycles lasting 2 weeks).

Total duration of the study: 24 months.

Number of Subjects:

Approximately 38 subjects will be enrolled on study:

- First stage:12 patients enrolled

If 1 or 0 responses were observed, the trial had to be terminated:

- Second stage: an additional of 23 patients were to be enrolled. If 5 or less responses were observed in 35 patients, the combination would not be considered worthy of further study, while if 6 or more responses were observed, the combination would be considered sufficiently active to warrant further testing. Taking into account an invalidity rate of 5%, 38 patients will be needed for this step.

DETAILED DESCRIPTION:
A Phase II Study to evaluate activity and toxicity of Gemcitabine in Combination with Pemetrexed long term infusion in the Treatment of pretreated Metastatic Colorectal Cancer Patients

Study Design:

Multicenter, non randomized, open label phase II study designed to evaluate the efficacy and safety of Gemcitabine/Pemetrexed combination.

Study Duration

Enrollment period: 18 months. Treatment period: maximum for 24 weeks for each patient (12 cycles lasting 2 weeks).

Total duration of the study: 24 months.

Primary objective:

- objective response rate (ORR: CR+PR+SD)

Secondary objectives:

* safety profile of the drugs combination;
* time to progression (TTP) and overall survival (OS)

Number of Subjects:

Approximately 38 subjects will be enrolled on study:

- First stage:12 patients enrolled

If 1 or 0 responses were observed, the trial had to be terminated:

- Second stage: an additional of 23 patients were to be enrolled. If 5 or less responses were observed in 35 patients, the combination would not be considered worthy of further study, while if 6 or more responses were observed, the combination would be considered sufficiently active to warrant further testing. Taking into account an invalidity rate of 5%, 38 patients will be needed for this step.

Statistical Methodology:

A minimax two-stage Simon design will be employed. A 10% response will preclude further study, whereas a 30% response rate will indicate that further study would be warranted. Using α and β errors of 0.10 and 0.10, respectively, 12 patients will be enrolled in the first stage, and if 1 or 0 responses were observed, the trial had to be terminated. Otherwise, an additional of 23 patients were to be enrolled, and if 5 or less responses were observed in 35 patients, the combination would not be considered worthy of further study, while if 6 or more responses were observed, the combination would be considered sufficiently active to warrant further testing. Taking into account an invalidity rate of 5%, 38 patients will be needed for this step.

The first 6 enrolled patients will be closely controlled for safety and further patients will be enrolled only in absence of severe toxicity resulting in discontinuation 1 month after the first cycle of the six patients.

The primary analysis will be performed on the ITT (Intention To Treat) population. PFS and OS will be estimated by the Kaplan-Meier method. The HR for PFS and OS will be estimated according to the Cox model, with its relative 95% confidence.

A secondary analysis will be performed on the PP (per-protocol) population. The Overall Response Rate to study treatment will be reported on the ITT and PP population with 95% confidence interval. Results will be tabulated and not evaluable patients will be included as additional category.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic confirmed diagnosis of colorectal carcinoma with metastatic (STAGE IV) disease.
2. Measurable disease according to RECIST criteria
3. Prior chemotherapy for metastatic disease is required; prior regimens (in adjuvant oral advanced stage setting) must include 5fluorouracile, Oxaliplatin and Irinotecan if not contraindicated.
4. At least a 4-week interval between the last dose of chemotherapy and study registration.
5. Recovery from all prior treatment-related toxicities to CTC <= grade 1 (except alopecia)
6. Male or female, aged >= 18 years
7. Life expectancy of greater than 12 weeks.
8. ECOG performance status <= 2
9. Patients must have normal organ and marrow function as defined below:

   * leukocytes >=3,000/microL
   * absolute neutrophil count >=1,500/microL
   * hemoglobin >= 9 g/dl
   * platelets >=100,000/microL
   * serum total bilirubin <= 1.5 X institutional upper limit of normal
   * AST(SGOT)/ALT(SGPT) <= 2.5 X institutional upper limit of normal (<= 5 times the upper institutional limits of normal if hepatic metastases are present)
   * serum creatinine <= 1.5 times the institutional upper limits of normal
   * Creatinine Clearance > 45 ml/min
10. The effects of Gemcitabine and Pemetrexed on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because therapeutic agents used in this trial are known to be teratogenic, female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception (hormonal or barrier method of birth control; abstinence) during the study and for 3 months thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. Participant is willing and able to give informed consent for participation in the study. Voluntary signed and dated written informed consent form in accordance with regulatory and institutional guidelines obtained before the performance of any protocol-related procedures not part of normal patient care.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
3. Previous treatment with Gemcitabine or Pemetrexed.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Gemcitabine and/or Pemetrexed or other agents used in the study
5. Patients with active brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
6. Past or current history of neoplasm other than colorectal carcinoma with a disease-free interval of less than 5 years, except for non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Inability to interrupt aspirin or other non-steroidal anti-inflammatory agents 2 days before, the day of, and 2 days after the dose of pemetrexed single agent or pemetrexed plus carboplatin.
9. HIV-positivity, whether or not symptomatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Determination of the objective response rate (ORR: CR (complete response) +PR (partial response) +SD (stable disease)) of treated patients according to RECIST criteria

SECONDARY OUTCOMES:
safety profile of study treatment | 2 years
  Assessment of safety profile of study drug combination in patients treated: report of Adverse Events according to the The NCI's Common Toxicity Criteria version 4.0
Time to Progression (TTP) | 2 years
  Determination of Time to Progression (TTP) of treated patients
Overall Survival (OS) | 2 years
  Determination of Overall Survival (OS) of treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luca Frassineti, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (1):
- UO Oncologia Medica IRCCS IRST, Meldola (FC), FC, Italy

REFERENCES:
- [Derived] Passardi A, Fanini F, Turci L, Foca F, Rosetti P, Ruscelli S, Casadei Gardini A, Valgiusti M, Dazzi C, Marangolo M. Prolonged Pemetrexed Infusion Plus Gemcitabine in Refractory Metastatic Colorectal Cancer: Preclinical Rationale and Phase II Study Results. Oncologist. 2017 Aug;22(8):886-e79. doi: 10.1634/theoncologist.2017-0206. Epub 2017 Jun 7. PMID 28592624